CLINICAL TRIAL: NCT01697592
Title: A Phase III, Multicenter, Randomized, Placebo-controlled, Parallel-group, Double-blinded Study and Subsequent Open-label, Extension Study to Assess the Safety and Efficacy of Addition of MK-3102 in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy and Oral Antihyperglycemic Agent Monotherapy
Brief Title: Omarigliptin (MK-3102) Clinical Trial - Add-on to Oral Antihyperglycemic Agent Study in Japanese Participants With Type 2 Diabetes Mellitus (MK-3102-015)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-015; 132242 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Omarigliptin 25 mg/Sulfonylureas (SUs) (Phase A+B) (Experimental): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of SUs throughout the duration of the study.
  Interventions: Drug: Omarigliptin
- Omarigliptin 25 mg/Glinides (Phase A+B) (Experimental): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of glinides throughout the duration of the study.
  Interventions: Drug: Omarigliptin
- Omarigliptin 25 mg/biguanides (BGs) (Phase A+B) (Experimental): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of BGs throughout the duration of the study.
  Interventions: Drug: Omarigliptin
- Omarigliptin 25 mg/Thiazolidinediones (TZDs) (Phase A+B) (Experimental): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of TZDs throughout the duration of the study.
  Interventions: Drug: Omarigliptin
- Omarigliptin 25 mg/α-GIs (Phase A+B) (Experimental): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of α-glucosidase (α-GIs) inhibitors throughout the duration of the study.
  Interventions: Drug: Omarigliptin
- Placebo/SUs (Phase A) → Omarigliptin 25 mg/SUs (Phase B) (Placebo Comparator): Placebo matching omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg is administered once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of SUs throughout the duration of the study.
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to omarigliptin
- Placebo/Glinides (Phase A) → Omarigliptin 25 mg/Gln. (Phase B) (Placebo Comparator): Placebo matching omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg is administered once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of glinides throughout the duration of the study.
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to omarigliptin
- Placebo/BGs (Phase A) → Omarigliptin 25 mg/BGs (Phase B) (Placebo Comparator): Placebo matching omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg is administered once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of BGs throughout the duration of the study.
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to omarigliptin
- Placebo/TZDs (Phase A) → Omarigliptin 25 mg/TZDs (Phase B) (Placebo Comparator): Placebo matching omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg is administered once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of TZDs throughout the duration of the study.
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to omarigliptin
- Placebo/α-GIs (Phase A) → Omarigliptin 25 mg/α-GIs (Phase B) (Placebo Comparator): Placebo matching omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg is administered once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of α-GIs inhibitors throughout the duration of the study.
  Interventions: Drug: Omarigliptin; Drug: Matching placebo to omarigliptin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin (MK-3102) 25 mg capsule administered orally once weekly. Pre-study basal medications include: SUs (gliclazide, glibenclamide, or glimepiride); Glinides (nateglinide , mitiglinide, or repaglinide); BGs (metformin); TZDs (pioglitazone); and α-GIs (acarbose, voglibose, or miglitol).
Drug: Matching placebo to omarigliptin — Matching placebo to omarigliptin 25 mg capsule administered orally once weekly. Pre-study basal medications include: SUs (gliclazide, glibenclamide, or glimepiride); Glinides (nateglinide , mitiglinide, or repaglinide); BGs (metformin); TZDs (pioglitazone); and α-GIs (acarbose, voglibose, or miglitol).
  Arms: Placebo/BGs (Phase A) → Omarigliptin 25 mg/BGs (Phase B); Placebo/Glinides (Phase A) → Omarigliptin 25 mg/Gln. (Phase B); Placebo/SUs (Phase A) → Omarigliptin 25 mg/SUs (Phase B); Placebo/TZDs (Phase A) → Omarigliptin 25 mg/TZDs (Phase B); Placebo/α-GIs (Phase A) → Omarigliptin 25 mg/α-GIs (Phase B)

SUMMARY:
This study will examine the safety and efficacy of the addition of omarigliptin in Japanese participants with type 2 diabetes mellitus who have inadequate glycemic control on diet/exercise therapy and oral antihyperglycemic agent monotherapy.

DETAILED DESCRIPTION:
The treatment period is composed of a 24-week double-blind period (Phase A) and a 28-week open-label period (Phase B). During Phase A, participants will received either omarigliptin 25 mg or a matching placebo. During Phase, B all participants will receive omarigliptin 25 mg. All participants will remain on a stable dose and administration of a single oral antihyperglycemic basal medication.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Has inadequate glycemic control on diet/exercise therapy and oral antihyperglycemic agent monotherapy

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of any of the following medications: Thiazolidinediones (TZD) (for participants whose basal medication is not TZD) and/or insulin within 12 weeks prior to study participation, omarigliptin anytime

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2014-05-08 (Actual); Study Completion 2014-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gantz I, Okamoto T, Ito Y, Sato A, Okuyama K, O'Neill EA, Engel SS, Lai E; Omarigliptin Study 015 Group. A Randomized, Placebo-Controlled Trial Evaluating the Safety and Efficacy of Adding Omarigliptin to Antihyperglycemic Therapies in Japanese Patients with Type 2 Diabetes and Inadequate Glycemic Control. Diabetes Ther. 2017 Aug;8(4):793-810. doi: 10.1007/s13300-017-0270-7. Epub 2017 Jun 6. PMID 28589493
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/study.html?id=3102-015&kw=3102-015&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-seven sites in Japan received IRB approval and were shipped clinical supplies in this study and randomized at least one participant. A total of 772 participants were screened of which 187 participants were excluded. The most common reason for participants not being randomized was screen failure (meeting exclusionary laboratory values).
Pre-assignment Details: In Phase A, participants were randomized to receive either omarigliptin (MK-3102) 25 mg once weekly or placebo for 24 weeks in a blinded manner. In Phase B, all participants received open-label omarigliptin 25 mg once weekly for 28 weeks.
Groups:
- Omarigliptin 25 mg/Sulfonylureas (SU) (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of SU throughout the duration of the study.
- Omarigliptin 25 mg/Glinides (Gln) (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Omarigliptin 25 mg/Biguanides (BG) (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of BG throughout the duration of the study.
- Omarigliptin 25 mg/Thiazolidinediones (TZD) (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Omarigliptin 25 mg/α-GI (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of α-glucosidase (α-GI) throughout the duration of the study.
- Placebo/SU (Phase A) Switching to Omari. 25 mg/SU (Phase B): Placebo to omarigliptin (omari.)administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of SU throughout the duration of the study.
- Placebo/Gln. (Phase A) Switching to Omari. 25 mg/Gln (Phase B): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Placebo/BG (Phase A) Switching to Omari. 25 mg/BG (Phase B): Placebo to Omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of BG. throughout the duration of the study.
- Placebo/TZD (Phase A) Switching to Omari. 25 mg/TZ (Phase B): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Placebo/α-GI (Phase A) Switching to Omari. 25 mg/α-GI (Ph. B): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of α-GI throughout the duration of the study.
Period: Phase A (Up to 24 Weeks)
Arm/Group | Omarigliptin 25 mg/Sulfonylureas (SU) (Phase A+B) | Omarigliptin 25 mg/Glinides (Gln) (Phase A+B) | Omarigliptin 25 mg/Biguanides (BG) (Phase A+B) | Omarigliptin 25 mg/Thiazolidinediones (TZD) (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Placebo/SU (Phase A) Switching to Omari. 25 mg/SU (Phase B) | Placebo/Gln. (Phase A) Switching to Omari. 25 mg/Gln (Phase B) | Placebo/BG (Phase A) Switching to Omari. 25 mg/BG (Phase B) | Placebo/TZD (Phase A) Switching to Omari. 25 mg/TZ (Phase B) | Placebo/α-GI (Phase A) Switching to Omari. 25 mg/α-GI (Ph. B)
Started | 126 | 65 | 66 | 65 | 67 | 63 | 34 | 33 | 34 | 32
Completed | 123 | 62 | 65 | 63 | 67 | 62 | 32 | 33 | 34 | 30
Not Completed | 3 | 3 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Period: Phase B (Week 25 to Week 52)
Arm/Group | Omarigliptin 25 mg/Sulfonylureas (SU) (Phase A+B) | Omarigliptin 25 mg/Glinides (Gln) (Phase A+B) | Omarigliptin 25 mg/Biguanides (BG) (Phase A+B) | Omarigliptin 25 mg/Thiazolidinediones (TZD) (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Placebo/SU (Phase A) Switching to Omari. 25 mg/SU (Phase B) | Placebo/Gln. (Phase A) Switching to Omari. 25 mg/Gln (Phase B) | Placebo/BG (Phase A) Switching to Omari. 25 mg/BG (Phase B) | Placebo/TZD (Phase A) Switching to Omari. 25 mg/TZ (Phase B) | Placebo/α-GI (Phase A) Switching to Omari. 25 mg/α-GI (Ph. B)
Started | 123 | 62 | 65 | 63 | 67 | 62 | 32 | 33 | 34 | 30
Completed | 118 | 61 | 64 | 60 | 67 | 60 | 31 | 32 | 32 | 30
Not Completed | 5 | 1 | 1 | 3 | 0 | 2 | 1 | 1 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Omarigliptin 25 mg/SU (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of SU throughout the duration of the study.
- Omarigliptin 25 mg/Gln (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Omarigliptin 25 mg/BG (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of BG throughout the duration of the study.
- Omarigliptin 25 mg/TZD (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Omarigliptin 25 mg/α-GI (Phase A+B): Omarigliptin 25 mg administered orally once weekly for 52 weeks (24 weeks during Phase A and 28 weeks during Phase B). Participants continued pre-study basal medication of α-GI throughout the duration of the study.
- Placebo/Gln (Phase A) Switching to Omari. 25 mg/Gln (Ph. B): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Placebo/BG (Phase A) Switching to Omari. 25 mg/BG (Phase B): Placebo to Omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of BG throughout the duration of the study.
- Placebo/TZD (Phase A) Switching to Omari. 25 mg/TZD (Phase B): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Omarigliptin 25 mg administered orally once weekly for 28 weeks during Phase B. Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 25 mg/SU (Phase A+B) | Omarigliptin 25 mg/Gln (Phase A+B) | Omarigliptin 25 mg/BG (Phase A+B) | Omarigliptin 25 mg/TZD (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Placebo/SU (Phase A) Switching to Omari. 25 mg/SU (Phase B) | Placebo/Gln (Phase A) Switching to Omari. 25 mg/Gln (Ph. B) | Placebo/BG (Phase A) Switching to Omari. 25 mg/BG (Phase B) | Placebo/TZD (Phase A) Switching to Omari. 25 mg/TZD (Phase B) | Placebo/α-GI (Phase A) Switching to Omari. 25 mg/α-GI (Ph. B) | Total
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 63 | 34 | 33 | 34 | 32 | 585
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (9) | 59 (11) | 59 (9) | 61 (10) | 61 (11) | 63 (11) | 61 (10) | 57 (9) | 61 (9) | 61 (11) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 19 | 20 | 23 | 21 | 18 | 7 | 10 | 7 | 9 | 169
  Male | 91 | 46 | 46 | 42 | 46 | 45 | 27 | 23 | 27 | 23 | 416

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event Excluding Data After Glycemic Rescue During Phase A
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure. Glycemic rescue criteria were: fasting plasma glucose (FPG) of >240 mg/dL, 2 times, (Week 4 to Week 24) and after Week 24, FPG >200 mg/dL, 2 times. Glycemic rescue was achieved through up-titration of basal medication (1st rescue) and through the use of metformin or glimepiride (2nd rescue).
Time Frame: Up to 24 weeks
Population: All Subjects as Treated (ASaT) population, defined as all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the ASaT population.
Measure: Number; unit: Percentage of participants
Groups:
- Omarigliptin 25 mg/SU (Phase A): Omarigliptin 25 mg administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of SU throughout the duration of the study.
- Omarigliptin 25 mg/Gln (Phase A): Omarigliptin 25 mg administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Omarigliptin 25 mg/BG (Phase A): Omarigliptin 25 mg administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of BG throughout the duration of the study.
- Omarigliptin 25 mg/TZD (Phase A): Omarigliptin 25 mg administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Omarigliptin 25 mg/α-GI (Phase A): Omarigliptin 25 mg administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of α-GI throughout the duration of the study.
- Placebo/SU (Phase A): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of SU throughout the duration of the study.
- Placebo/Gln. (Phase A): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Placebo/BG (Phase A): Placebo to Omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of BG throughout the duration of the study.
- Placebo/TZD (Phase A): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Placebo/α-GI (Phase A): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of α-GI throughout the duration of the study.
Arm/Group | Omarigliptin 25 mg/SU (Phase A) | Omarigliptin 25 mg/Gln (Phase A) | Omarigliptin 25 mg/BG (Phase A) | Omarigliptin 25 mg/TZD (Phase A) | Omarigliptin 25 mg/α-GI (Phase A) | Placebo/SU (Phase A) | Placebo/Gln. (Phase A) | Placebo/BG (Phase A) | Placebo/TZD (Phase A) | Placebo/α-GI (Phase A)
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 63 | 34 | 33 | 34 | 32
Percentage of participants | 59.5 | 53.8 | 54.5 | 60.0 | 50.7 | 60.3 | 52.9 | 63.6 | 52.9 | 53.1

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event Excluding Data After Glycemic Rescue During the Overall Study
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure. Glycemic rescue criteria were: fasting plasma glucose (FPG) of >240 mg/dL, 2 times, (Week 4 to Week 24) and after Week 24, FPG >200 mg/dL, 2 times. Glycemic rescue was achieved through up-titration of basal medication (1st rescue) and through the use of metformin or glimepiride (2nd rescue). These results represent the accrual of events over different treatment intervals: 52 weeks, Omarigliptin (Phase A+B) group, defined as the double-blind period and open-label extension period versus 28 weeks for the placebo switching to Omarigliptin group defined as the open-label extension period only.
Time Frame: Up to 52 weeks
Population: The ASaT population was all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data. Data was unavailable for 5 participants who discontinued from the study in the placebo arm in Phase A.
Measure: Number; unit: Percentage of participants
Groups:
- Omarigliptin 25mg/SU (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo.
  Participants continued prestudy basal medication of SU throughout the duration of the study.
- Omarigliptin 25mg/Gln (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo.
  Participants continued pre-study basal medication of Gln throughout the duration of the study.
- Omarigliptin 25mg/BG (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo. Participants continued pre-study basal medication of BG throughout the duration of the study.
- Omarigliptin 25mg/TZD (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo. Participants continued pre-study basal medication of TZD throughout the duration of the study.
- Omarigliptin 25mg/α-GI (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo. Participants continued pre-study basal medication of α-GI throughout the duration of the study.
Arm/Group | Omarigliptin 25 mg/SU (Phase A+B) | Omarigliptin 25 mg/Gln (Phase A+B) | Omarigliptin 25 mg/BG (Phase A+B) | Omarigliptin 25 mg/TZD (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Omarigliptin 25mg/SU (Phase B) | Omarigliptin 25mg/Gln (Phase B) | Omarigliptin 25mg/BG (Phase B) | Omarigliptin 25mg/TZD (Phase B) | Omarigliptin 25mg/α-GI (Phase B)
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 62 | 32 | 33 | 34 | 30
Percentage of participants | 76.2 | 75.4 | 80.3 | 84.6 | 68.7 | 56.5 | 59.4 | 66.7 | 58.8 | 53.3

3. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event During Phase A
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 24 weeks
Population: The ASaT population was defined as all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data using the ASaT population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Omarigliptin 25 mg/SU (Phase A) | Omarigliptin 25 mg/Gln (Phase A) | Omarigliptin 25 mg/BG (Phase A) | Omarigliptin 25 mg/TZD (Phase A) | Omarigliptin 25 mg/α-GI (Phase A) | Placebo/SU (Phase A) | Placebo/Gln. (Phase A) | Placebo/BG (Phase A) | Placebo/TZD (Phase A) | Placebo/α-GI (Phase A)
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 63 | 34 | 33 | 34 | 32
Percentage of Participants | 0 | 3.1 | 0 | 3.1 | 0 | 0 | 2.9 | 0 | 0 | 3.1

4. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event During the Overall Study
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Omarigliptin 25mg/BG (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo. Participants continued pre-study basal medication of BG. throughout the duration of the study.
Arm/Group | Omarigliptin 25 mg/SU (Phase A+B) | Omarigliptin 25 mg/Gln (Phase A) | Omarigliptin 25 mg/BG (Phase A+B) | Omarigliptin 25 mg/TZD (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Omarigliptin 25mg/SU (Phase B) | Omarigliptin 25mg/Gln (Phase B) | Omarigliptin 25mg/BG (Phase B) | Omarigliptin 25mg/TZD (Phase B) | Omarigliptin 25mg/α-GI (Phase B)
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 62 | 32 | 33 | 34 | 30
Percentage of participants | 0.8 | 4.6 | 1.5 | 6.2 | 0 | 1.6 | 0 | 0 | 2.9 | 0

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24
Description: HbA1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%). Thus, this change from baseline reflects the Week 24 HbA1c minus the Week 0 HbA1c.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS), comprised of all participants who received at least one study drug and have a baseline or post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent HbA1C
Groups:
- Placebo/Gln. (Phase A): Placebo to omarigliptin administered orally once weekly for 24 weeks during Phase A. Participants continued pre-study basal medication of Gln. throughout the duration of the study.
Arm/Group | Omarigliptin 25 mg/SU (Phase A) | Omarigliptin 25 mg/Gln (Phase A) | Omarigliptin 25 mg/BG (Phase A) | Omarigliptin 25 mg/TZD (Phase A) | Omarigliptin 25 mg/α-GI (Phase A) | Placebo/SU (Phase A) | Placebo/Gln. (Phase A) | Placebo/BG (Phase A) | Placebo/TZD (Phase A) | Placebo/α-GI (Phase A)
Number analyzed (Participants) | 126 | 65 | 66 | 65 | 67 | 63 | 34 | 33 | 34 | 32
Percent HbA1C | -0.84 [-0.94 to -0.73] | -0.68 [-0.89 to -0.48] | -0.94 [-1.10 to -0.78] | -0.88 [-1.04 to -0.73] | -0.74 [-0.89 to -0.59] | 0.09 [-0.06 to 0.24] | 0.30 [-0.04 to 0.64] | -0.02 [-0.35 to 0.31] | 0.28 [0.03 to 0.53] | 0.06 [-0.16 to 0.28]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg/SU (Phase A) vs Placebo/SU (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Constrained longitudinal data analysis with terms for treatment, basal AHA medication, prior AHA therapy status except for basal medication, and time; Difference in the least squares means = -0.93, 95% CI 2-sided [-1.10 to -0.75]
Statistical Analysis 2: Comparison: Omarigliptin 25 mg/Gln (Phase A) vs Placebo/Gln. (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 5, analysis 1]; Difference in the least squares means = -0.98, 95% CI 2-sided [-1.37 to -0.60]
Statistical Analysis 3: Comparison: Omarigliptin 25 mg/BG (Phase A) vs Placebo/BG (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 5, analysis 1]; Difference in the least squares means = -0.92, 95% CI 2-sided [-1.29 to -0.56]
Statistical Analysis 4: Comparison: Omarigliptin 25 mg/TZD (Phase A) vs Placebo/TZD (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 5, analysis 1]; Difference in the least squares means = -1.16, 95% CI 2-sided [-1.45 to -0.88]
Statistical Analysis 5: Comparison: Omarigliptin 25 mg/α-GI (Phase A) vs Placebo/α-GI (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 5, analysis 1]; Difference in the least squares means = -0.80, 95% CI 2-sided [-1.06 to -0.54]

ADVERSE EVENTS:
Time Frame: Phase A (up to 24 weeks), Phase A+B (up to 52 weeks). Phase B (Up to 28 weeks [Week 25 to 52])
Description: The ASaT Population was used for this analysis. AEs occuring after glycemic rescue were included in the analysis of SAEs but not for Non-SAEs. 5 participants in the placebo arm discontinued from the study in Phase A. The AEs for the various placebo arms were grouped into 1 placebo arm regardless of the antihyperglycemic basal medication received.
Groups:
- Placebo/ABM (Phase A): Placebo to omargliptin administered orally once weekly for 24 weeks during Phase A. Participants continued any pre-study basal medication (ABM)throughout the duration of the study.
- Omarigliptin 25mg/ABM (Phase B): Omarigliptin 25mg administered orally once weekly for 28 weeks during Phase B after switching from placebo.
  Participants continued any prestudy basal medications throughout the duration of the study.
Arm/Group | Omarigliptin 25 mg/SU (Phase A) | Omarigliptin 25 mg/Gln (Phase A) | Omarigliptin 25 mg/BG (Phase A) | Omarigliptin 25 mg/TZD (Phase A) | Omarigliptin 25 mg/α-GI (Phase A) | Placebo/ABM (Phase A) | Omarigliptin 25 mg/SU (Phase A+B) | Omarigliptin 25 mg/Gln (Phase A+B) | Omarigliptin 25 mg/BG (Phase A+B) | Omarigliptin 25 mg/TZD (Phase A+B) | Omarigliptin 25 mg/α-GI (Phase A+B) | Omarigliptin 25mg/ABM (Phase B)
Serious Adverse Events (participants affected / at risk) | 3/126 | 1/65 | 1/66 | 4/65 | 0/67 | 4/196 | 6/126 | 3/65 | 2/66 | 4/65 | 1/67 | 7/191
Other Adverse Events (participants affected / at risk) | 33/126 | 19/65 | 22/66 | 18/65 | 19/67 | 62/196 | 58/126 | 29/65 | 33/66 | 30/65 | 26/67 | 60/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg/SU (Phase A) (N=126) | Omarigliptin 25 mg/Gln (Phase A) (N=65) | Omarigliptin 25 mg/BG (Phase A) (N=66) | Omarigliptin 25 mg/TZD (Phase A) (N=65) | Omarigliptin 25 mg/α-GI (Phase A) (N=67) | Placebo/ABM (Phase A) (N=196) | Omarigliptin 25 mg/SU (Phase A+B) (N=126) | Omarigliptin 25 mg/Gln (Phase A+B) (N=65) | Omarigliptin 25 mg/BG (Phase A+B) (N=66) | Omarigliptin 25 mg/TZD (Phase A+B) (N=65) | Omarigliptin 25 mg/α-GI (Phase A+B) (N=67) | Omarigliptin 25mg/ABM (Phase B) (N=191)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg/SU (Phase A) (N=126) | Omarigliptin 25 mg/Gln (Phase A) (N=65) | Omarigliptin 25 mg/BG (Phase A) (N=66) | Omarigliptin 25 mg/TZD (Phase A) (N=65) | Omarigliptin 25 mg/α-GI (Phase A) (N=67) | Placebo/ABM (Phase A) (N=196) | Omarigliptin 25 mg/SU (Phase A+B) (N=126) | Omarigliptin 25 mg/Gln (Phase A+B) (N=65) | Omarigliptin 25 mg/BG (Phase A+B) (N=66) | Omarigliptin 25 mg/TZD (Phase A+B) (N=65) | Omarigliptin 25 mg/α-GI (Phase A+B) (N=67) | Omarigliptin 25mg/ABM (Phase B) (N=191)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 15 (17) | 14 (16) | 11 (14) | 11 (13) | 13 (14) | 44 (49) | 34 (44) | 23 (30) | 24 (34) | 19 (29) | 19 (25) | 36 (44)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (10) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 3 (7) | 11 (14) | 2 (3) | 3 (7) | 2 (2) | 0 (0) | 6 (7)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 7 (8) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 10 (10) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 7 (10)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 6 (6) | 4 (4) | 4 (4) | 5 (6) | 4 (4) | 10 (11)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.